CLINICAL TRIAL: NCT01879332
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Multiple Ascending Dose Study of the Safety and Pharmacokinetics of Eslicarbazepine Acetate in Adult Healthy Volunteers
Brief Title: A Sequential Multiple Ascending Dose Study of the Safety and Pharmacokinetics of Eslicarbazepine Acetate in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-118
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
Keywords: Anticonvulsant
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo tablets for oral administration
  Interventions: Drug: Placebo
- BIA 2-093 3000 mg once daily (Experimental): Subjects in Cohort 2 received a dose of 3000 mg once daily (5 x 600 mg eslicarbazepine acetate tablets)
  Interventions: Drug: BIA 2-093 3000 mg once daily
- BIA 2-093 3600 mg once daily (Experimental): Subjects in Cohort 1 received a dose of 3600 mg once daily (6 x 600 mg eslicarbazepine acetate tablets)
  Interventions: Drug: BIA 2-093 3600 mg once daily

INTERVENTIONS:
Drug: Placebo — Matching placebo tablets for oral administration
  Other Names: sugar pills
  Arms: Placebo
Drug: BIA 2-093 3000 mg once daily — Eslicarbazepine acetate 600 mg tablets for oral administration
  Other Names: eslicarbazepine acetate
  Arms: BIA 2-093 3000 mg once daily
Drug: BIA 2-093 3600 mg once daily — Eslicarbazepine acetate 600 mg tablets for oral administration
  Other Names: Eslicarbazepine acetate
  Arms: BIA 2-093 3600 mg once daily

SUMMARY:
Randomized, double-blind, placebo-controlled, sequential multiple ascending dose study to determine a maximum tolerated dose

DETAILED DESCRIPTION:
This study was designed as a randomized, double-blind, placebo-controlled, sequential multiple ascending dose study to assess the safety and pharmacokinetics of supratherapeutic doses of eslicarbazepine acetate in 32 healthy adult male and female subjects, with 8 subjects per treatment group. In each study group, subjects were to receive single doses of eslicarbazepine acetate or placebo once daily for 5 days.

A series of screening evaluations was performed within a 21-day period prior to the first dose of study medication in order to determine the eligibility of prospective study participants for the trial. Eligible subjects reported to the clinic on Day -1 prior to study medication administration and remained in the clinic until clinic discharge on Day 7. Plasma and urine samples were collected throughout the study to determine the pharmacokinetics of eslicarbazepine acetate and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 18 to 45 years of age. Women were required to be postmenopausal (more than 12 months since last period); surgically sterile (hysterectomy or tubal ligation at least 6 months prior to enrollment); using an intrauterine device; or double barrier (i.e. diaphragm or spermicide plus male condom) non-hormonal contraceptive therapy for the duration of the trial. Female subjects were required to have a negative pregnancy test at screening and upon check-in to the study facility.
* BMI within the range of 18-30 kg/m2.
* Ability to communicate effectively with the study personnel.
* No significant disease or abnormal laboratory values as determined by medical history, physical examination or laboratory evaluations, conducted at the screening visit and on admission to the clinic.
* Normal 12-lead electrocardiogram, without any clinically significant abnormalities of rate, rhythm or conduction.
* Nonsmokers defined as not having smoked in the past 6 months.
* Subjects were to be adequately informed of the nature and risks of the study and were required to provide written informed consent prior to study entry.

Exclusion Criteria:

* Known hypersensitivity or allergy to eslicarbazepine acetate or related compounds such as carbamazepine, oxcarbazepine, or licarbazepine.
* Women who were pregnant or breast feeding.
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, had the potential to compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that could interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk.
* A sustained supine systolic blood pressure > 140 mmHg or <100mmHg or a diastolic blood pressure > 95 mmHg at screening or baseline.
* A resting ECG heart rate of <50 bpm or >100 bpm.
* An abnormal screening ECG indicating a second- or third-degree AV block, or one or more of the following: QRS > 110 milliseconds (msec), QTc (Fridericia correction) > 450 msec, PR interval > 240 msec. Any rhythm other than sinus rhythm, which was interpreted by the Investigator to be clinically significant.
* The presence of abnormal laboratory values which were considered clinically significant.
* Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti HCV, Hepatitis C Antibody), or HIV (anti-HIV 1 or 2).
* Receipt of an investigational drug within a period of 30 days prior to enrollment in the study.
* Receipt of any drug therapy, including hormonal contraceptives, within 2 weeks prior to administration of the first dose of any study-related treatment. This exclusion was extended to 4 weeks for any drugs known to induce or inhibit hepatic drug metabolism.
* Consumption of alcohol within 48 hours prior to dose administration or during any in-patient period.
* A positive urine drug screen including ethanol, cocaine, THC, barbiturates, amphetamines, benzodiazepines, and opiates.
* Any history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction.
* A history of difficulty with donating blood.
* Donation of blood or blood products within 45 days prior to enrollment.
* Subjects with, or with a history of, additional risk factors for Torsades de Points (e.g., heart failure, hypokalemia), or a family history of long QT syndrome or family history of sudden death.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Phase OneTM, Miramar, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIA 2-093 3000 mg Once Daily | BIA 2-093 3600 mg Once Daily | Placebo
Started | 6 | 6 | 4
Completed | 0 | 0 | 0
Not Completed | 6 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BIA 2-093 3000 mg Once Daily | BIA 2-093 3600 mg Once Daily | Total
Number analyzed (Participants) | 4 | 6 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 6 | 16
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4 | 8
  Male | 4 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Reported
Description: Safety was evaluated through the recording and monitoring of adverse events
Time Frame: 2 days
Measure: Number; unit: Number of adverse events reported
Arm/Group | BIA 2-093 3000 mg Once Daily | BIA 2-093 3600 mg Once Daily | Placebo
Number analyzed (Participants) | 6 | 6 | 4
Number of adverse events reported
  Nervous system AE | 6 | 6 | 1
  Gastrointestinal AE | 5 | 4 | 1
  General and Administration Site Conditions AE | 4 | 1 | 0
  Eye AE | 1 | 1 | 0
  Skin and Subcutaneous Tissue AE | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | BIA 2-093 3000 mg Once Daily | BIA 2-093 3600 mg Once Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 3000 mg Once Daily (N=6) | BIA 2-093 3600 mg Once Daily (N=6) | Placebo (N=4)
Dizziness (Nervous system disorders) | 5 | 5 | 1
Somnolence (Nervous system disorders) | 0 | 4 | 1
Headache (Nervous system disorders) | 3 | 0 | 0
Paraesthesia Oral (Nervous system disorders) | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 4 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other